CLINICAL TRIAL: NCT00922064
Title: Effects of Electroconvulsive Therapy on Serotonin-1A Receptor Binding in Major Depression
Brief Title: Effects of Electroconvulsive Therapy (ECT) on Serotonin-1A Receptor Binding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, A/Prof. PD Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EKT-20090219 Version 1.3; MUW EC No. 556/2008
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Unipolar Depression
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ECT (Experimental)
  Interventions: Procedure: ECT

INTERVENTIONS:
Procedure: ECT — ECT series consisting of 6 to 14 ECTs

SUMMARY:
In treatment-resistant depression, electroconvulsive therapy (ECT) has been shown to effectively reduce depressive symptoms, though the underlying neurobiological mechanism is still unclear. The serotonergic system, and in particular the inhibitory serotonin-1A (5-HT1A) receptor, appears to be significantly involved in the effectiveness of ECT. The aim of the study is to assess the effects of ECT on the 5-HT1A receptor binding potential (BPND) and distribution in humans in vivo using positron emission tomography (PET) and the radioligand [carbonyl-11C]WAY-100635.

12 patients suffering from severe, therapy-resistant unipolar depression will undergo 3 PET scans, two of these scans taking place before the ECT treatment, consisting of 6-14 ECTs, the third scan taking place after the ECT treatment.

This imaging study hypothesizes that upon completion of the ECT, the overall 5-HT1A receptor BPND in the brain of depressed patients will significantly change.

This study would be the first to demonstrate an effect of electroconvulsive therapy on the 5-HT1A receptor binding in humans in vivo. Given the involvement of the 5-HT1A receptor in the pathophysiology of mood disorders, the present study would be an important step towards a better understanding of antidepressant treatment and treatment response. By comparing treatment effect and the underlying biological mechanism, the study might help to identify biomarkers that distinguish patients who are likely to benefit from ECT from patients who will rather be non-responders. Finally, by investigating the role of the 5-HT1A receptor in ECT, is highly discussed relevance for antidepressant action will be further elucidated and might prepare the ground for new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 - 65 years
* ICD-10 diagnosis of severe unipolar depression (ICD-10: F32.2, F32.3; F33.2, F33.3)
* A score of 23 or greater on the 17-item HAM-D
* Signed informed consent form
* Negative urine pregnancy test in women at the screening visit and at PET days
* Antidepressive and antipsychotic medication in a steady state for at least 10 days prior to inclusion
* Anesthesiological approval for ECT

Exclusion Criteria:

* Concomitant major internistic or neurological illness
* Clinically relevant abnormalities on a general physical examination and routine laboratory screening
* Current substance abuse, addiction
* Current or past history of schizophrenia or schizoaffective disorder
* Exposure to artificial radiation as volunteer in clinical studies within 10 years prior to inclusion into the present study
* Previous treatments with electroconvulsive therapy
* Treatment (< 1 months before screening) with the following drugs: Aripiprazole, Risperidone, Ziprasidone, Clozapine, Chlorpromazine, Amitryptyline, Nefazodone, Trazodone, Buspirone, Pindolol, Penbutolol, Tertatolol, Alprenolol, Quetiapine
* Investigations using PET or SPECT within 10 years prior to the inclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
serotonin-1A receptor binding potential | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Frey, MD, Principal Investigator — Medical University of Vienna, Dept. of Psychiatry and Psychotherapy
Locations (1):
- Medical University of Vienna, Dept. of Psychiatry and Psychotherapy, Vienna, Vienna, Austria